CLINICAL TRIAL: NCT00194649
Title: Glycosphingolipid Inhibition and Spermatogenesis in Man: A Pilot Study
Brief Title: Glycosphingolipid Inhibition and Spermatogenesis in Man: A Pilot Study (MIG 2)
Acronym: MIG-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: John K Amory, MD, MPH, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-3806-D; U54HD042454 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Contraception
Keywords: Glycosphingolipids (GSL)
MeSH Terms: interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 100 mg Miglustat BID (twice daily) for six weeks
  Interventions: Drug: Miglustat (Zavesca)

INTERVENTIONS:
Drug: Miglustat (Zavesca) — 100 mg Miglustat BID (twice daily) for six weeks
  Other Names: Zavseca

SUMMARY:
The purpose of this research study is to help in the development of safe, effective and reversible male contraception. We are examining the impact of the drug Miglustat on sperm production in normal men.

We want to see if Miglustat will inhibit sperm production in men and act as a reversible male contraceptive, as a study in mice administered Miglustat showed a reversible inhibition of sperm production. We believe Miglustat may have some potential as a safe, reversible male contraceptive.

DETAILED DESCRIPTION:
Glycosphingolipids (GSL) are a main constituent of the sperm cell membrane in mammals. Male mice deficient in enzymes involved in GSL synthesis have severely impaired fertility and knockout mice are infertile. Recently, it was demonstrated that administration to mice of an inhibitor of ceramide-specific glycosyltransferase, the first step in the biosynthetic pathway of GSL formation, resulted in reversible infertility without discernable adverse side effects. This inhibitor was Miglustat, which is an alkylated imino sugar. The impact of Miglustat therapy on human spermatogenesis is unknown. If the effects on sperm morphology and motility are similar to those observed in mice, Miglustat or other GSL inhibitors might have potential utility as non-hormonal male contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, normal lab test

Exclusion Criteria:

* Abnormal lab test, history or evidence of significant chronic or acute medical illness, previous or current ethanol or anabolic steroid abuse.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-06; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The impact of GSL inhibition on human spermatogenesis, if impairment is seen with Miglustat administration, larger contraceptive efficacy studies of Miglustat or other inhibitors of GSL's will be performed. | 3 months

SECONDARY OUTCOMES:
Safety | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John Amory, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Takamiya K, Yamamoto A, Furukawa K, Zhao J, Fukumoto S, Yamashiro S, Okada M, Haraguchi M, Shin M, Kishikawa M, Shiku H, Aizawa S, Furukawa K. Complex gangliosides are essential in spermatogenesis of mice: possible roles in the transport of testosterone. Proc Natl Acad Sci U S A. 1998 Oct 13;95(21):12147-52. doi: 10.1073/pnas.95.21.12147. PMID 9770454
- [Background] Ritter G, Krause W, Geyer R, Stirm S, Wiegandt H. Glycosphingolipid composition of human semen. Arch Biochem Biophys. 1987 Sep;257(2):370-8. doi: 10.1016/0003-9861(87)90579-0. PMID 3662530
- [Background] Fujimoto H, Tadano-Aritomi K, Tokumasu A, Ito K, Hikita T, Suzuki K, Ishizuka I. Requirement of seminolipid in spermatogenesis revealed by UDP-galactose: Ceramide galactosyltransferase-deficient mice. J Biol Chem. 2000 Jul 28;275(30):22623-6. doi: 10.1074/jbc.C000200200. PMID 10801776
- [Background] Honke K, Hirahara Y, Dupree J, Suzuki K, Popko B, Fukushima K, Fukushima J, Nagasawa T, Yoshida N, Wada Y, Taniguchi N. Paranodal junction formation and spermatogenesis require sulfoglycolipids. Proc Natl Acad Sci U S A. 2002 Apr 2;99(7):4227-32. doi: 10.1073/pnas.032068299. Epub 2002 Mar 26. PMID 11917099
- [Background] Platt FM, Neises GR, Karlsson GB, Dwek RA, Butters TD. N-butyldeoxygalactonojirimycin inhibits glycolipid biosynthesis but does not affect N-linked oligosaccharide processing. J Biol Chem. 1994 Oct 28;269(43):27108-14. PMID 7929454
- [Background] van der Spoel AC, Jeyakumar M, Butters TD, Charlton HM, Moore HD, Dwek RA, Platt FM. Reversible infertility in male mice after oral administration of alkylated imino sugars: a nonhormonal approach to male contraception. Proc Natl Acad Sci U S A. 2002 Dec 24;99(26):17173-8. doi: 10.1073/pnas.262586099. Epub 2002 Dec 11. PMID 12477936
- [Background] Beutler E. Gaucher disease. Curr Opin Hematol. 1997 Jan;4(1):19-23. doi: 10.1097/00062752-199704010-00004. PMID 9050375
- [Result] Amory JK, Muller CH, Page ST, Leifke E, Pagel ER, Bhandari A, Subramanyam B, Bone W, Radlmaier A, Bremner WJ. Miglustat has no apparent effect on spermatogenesis in normal men. Hum Reprod. 2007 Mar;22(3):702-7. doi: 10.1093/humrep/del414. Epub 2006 Oct 25. PMID 17067996